CLINICAL TRIAL: NCT02419300
Title: Value of Pelvic Ultrasonography and Colour Doppler in Diagnosing Retained Placental Fragments After Mid Trimester Miscarriage
Brief Title: Could Colour Dopper Improve the Diagnosis of Retained Placental Fragments After Second Trimester Miscarriage ?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed El Kotb Abdel Fattah, lecturer, Ain Shams University
Other Study IDs: USDIA
Record Dates: First submitted 2015-04-10; First posted 2015-04-17 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Miscarriage
MeSH Terms: conditions — Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: ultrasoungraphy — pelvic ultrasonography and Doppler

SUMMARY:
Value of pelvi- abdominal ultrasound and Doppler in diagnosis of retained products of conception after second trimester miscarriage to select who will benefit from surgical evacuations or conservative management.

DETAILED DESCRIPTION:
This is a study for diagnostic accuracy test where all patients will undergo US and Doppler examination after second trimester miscarriage. Then all patients with endometrial mass on US will undergo colour Doppler then surgical evacuation and results of histopathology will be recorded.

Now, pathological examination of suction evacuation products is considered the gold standard so sensitivity, specificity, PPV and NPV of US and Doppler are the primary outcome

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy duration: early mid-trimester from 14 to 20 weeks
* Endometrial mass upon ultrasound examination after second trimesteric miscarriage

Exclusion Criteria:

* Uterine congenital anomaly
* Patients with signs of sepsis.
* Negative scan after second trimesteric miscarriage

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients visiting The Obstetrics department in Ain Shams University Hospital complaining of early second trimesteric abortion
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-03 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Sensitivity, specificity, PPV and NPV of Doppler in diagnosis of retained placental fragments after second trimester miscarriage | 60 minutes after delivery
  All patients with endometrial mass after spontineous or medical miscarriage will undergo colour Doppler examination within 1 hour of miscarriage

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Ain Shams University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes